CLINICAL TRIAL: NCT06269458
Title: The Effects of Mother-Baby Yoga and Baby Massage on Attachment and Sleep: A Randomized Crossover Pilot Study
Brief Title: The Effects of Mother-Baby Yoga and Baby Massage on Attachment and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ABU-001
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Newborn; Yoga; Mother-Infant Interaction; Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby Massage (Experimental): In the baby massage application, mothers were trained on baby massage and the massage applied by the mother to her baby was observed once. The baby massage video prepared by the researchers was shared with mothers. Baby massage application was performed 90 minutes after feeding and each application was performed at the same time. Mothers massaged their babies for 15 minutes three times a week for a month. The Massage Application Content included one minute face, two minutes chest, four minutes arm, two minutes abdominal, four minutes leg and two minutes back massage (Virgian and Setiawati, 2021; Yenigün 2020; Yılmaz, 2019). All mothers were called once a week by a researcher to provide counseling and follow-up of the process.
  At the end of four weeks, measurement tools were applied to all mothers and the groups were changed, massage was applied to the yoga group, and yoga intervention was applied to the massage group, as in the beginning of the research.
  Interventions: Behavioral: Baby Massage
- Mother-Baby Yoga (Experimental): The mothers in the Mother-Baby Yoga group were given a 10-minute training on mother-baby yoga before the application, and then a session was applied together. Mothers were asked to choose the most suitable time of day for themselves and the baby, to ensure that the baby was fed at least 45 minutes before yoga, and to practice yoga in a calm and dimly lit environment, listening to music or white noise of their choice. One yoga session lasted approximately 20 minutes. Mothers and their babies did mother-baby yoga three times a week for four weeks. Mother baby yoga content; Mood regulation: belly breathing, warm touch from the heart, chair pose, scoop hug, bukka bukka, vortex creation, lush falls one hand two hands, tiny stretches, here and now awareness and dolphin pose.
  Interventions: Behavioral: Monther-Baby Yoga

INTERVENTIONS:
Behavioral: Baby Massage — In the baby massage application, mothers were trained on baby massage and the massage applied by the mother to her baby was observed once. The baby massage video prepared by the researchers was shared with mothers. Mothers were informed about the importan
  Arms: Baby Massage
Behavioral: Monther-Baby Yoga — Mothers were asked to choose the most suitable time of day for themselves and the baby, to ensure that the baby was fed at least 45 minutes before yoga, and to practice yoga in a calm and dimly lit environment, listening to music or white noise of their choice. One yoga session lasted approximately 20 minutes. Mothers and their babies did mother-baby yoga three times a week for four weeks. Mothers were informed about the importance of having the same treatment room for each treatment. All mothers were called once a week by a researcher to provide counseling and follow-up of the process.
  At the end of four weeks, measurement tools were applied to all mothers and the groups were changed, massage was applied to the yoga group, and yoga intervention was applied to the massage group, as in the beginning of the research. At the end of four weeks, all mothers were evaluated for mother-infant attachment and the infant's sleep diary.
  Arms: Mother-Baby Yoga

SUMMARY:
Purpose: This study was conducted to examine the effects of mother-baby yoga and massage on mother-baby bonding and the baby's sleep.

Method: A randomised, crossover pilot study was conducted in the postpartum service of a hospital between January and November 2023, with 60 mothers and their babies in the postpartum period, 30 in each group. To the mothers and their babies included in the research, baby massage was applied to one group and mother-baby yoga was applied to the other. After four weeks, the groups' practices were changed. In the results of the research, characteristics related to attachment and sleep were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Babies in the first week of postpartum
* Healthy babies,
* Therm (37-40 W),
* The baby should be at normal birth weight (2500-4000gr),
* Mothers who know how to read and writ

Exclusion Criteria:

* Mothers with communication problems,
* Individuals whose mother or baby are monitored in intensive care after birth
* If the mother has a physical disability or any chronic disease (hypertension, diabetes mellitus, etc.),
* Psychological illness in the mother (major depression, psychosis, etc.),
* Pregnancy through assisted reproductive techniques,
* Mothers who are diagnosed with a sleep disorder and who have their babies treated for this reason.

Ages: 0 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Attachment | It was applied before and after the intervention (4 weeks).
  The Mother-Infant Attachment Scale developed by Taylor et al. was used to measure mother-infant attachment. The Turkish validity and reliability study of the scale was conducted by (Karakulak et al., 2016). The MIBS is designed to be administered from the first day after birth and allows the mother to express her feelings towards her baby with a single word. This scale, which can be easily and quickly administered by the mother or father alone, shows the relationship between the established bond and the mother's early mood.
Weight and Sleep | It was applied before and after the intervention (4 weeks).
  Sleep characteristics of the infants were assessed using a sleep diary form created by the researchers. The form included questions about the time of starting the bedtime routine, the time of going to bed, the number of nighttime awakenings, the duration of staying awake at night, the longest sleep time spent without waking up at night, the total sleep time at night, the number of daytime naps, and the total sleep time during the day (Ağapınar et al., 2023; Del-Ponte et al., 2020; Hanifarizani et al., 2020; Mrljak et al., 2022). The mothers were asked to write in this diary to be recorded for one day during the first and last week of the implementation process.

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya Bilim Üniversitesi, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study will be shared after it is published.